CLINICAL TRIAL: NCT05293080
Title: Early Treatment of Atrial Fibrillation for Stroke Prevention Trial in Acute STROKE
Acronym: EAST-STROKE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Heart & Vascular Center Hamburg, Department of Cardiology (Unknown); Department of Neurology, Royal Melbourne Hospital (Unknown); Melbourne Heart Centre, Royal Melbourne Hospital (Unknown); Hotchkiss Brain Institute, University of Calgary (Other); Department of Neurology and Neurosurgery, Brain Center, University Medical Center Utrecht (Unknown); UMC Utrecht (Other); Edinburgh Clinical Trials Unit, Cerebrovascular Research Group, Centre for Clinical Brain Sciences, University of Edinburgh (Unknown); Department of Cardiovascular Sciences, University of Leicester British Heart Foundation Cardiovascular Research Centre (Unknown); Institute of Medical Biometry and Epidemiology, University Medical Center Hamburg-Eppendorf (Unknown); CTC-NORTH (Unknown); Stroke Alliance for Europe (SAFE) (Unknown); Kompetenznetz Vorhofflimmern e.V. (AFNET) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EAST-STROKE
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation
Keywords: Acute ischemic stroke; Atrial fibrillation; Rhythm control; Ablation; Antiarrhythmic drugs
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early rhythm control therapy (Experimental): Patients with acute ischemic stroke and AF will receive either catheter ablation (mainly pulmonary vein isolation), or adequate antiarrhythmic drug therapy at an early time point. The initial therapy will be selected by the local investigator. In case of continuation or recurrence of AF, both modalities may be combined.
  Interventions: Other: Medical or interventional therapy for rhythm control in atrial fibrillation (antiarrhythmic drugs, ablation, electric cardio version)
- Usual care (Active Comparator): Patients with acute ischemic stroke and AF will receive usual care following the current ESC guidelines for AF treatment.
  Interventions: Other: Usual care for atrial fibrillation

INTERVENTIONS:
Other: Medical or interventional therapy for rhythm control in atrial fibrillation (antiarrhythmic drugs, ablation, electric cardio version) — Therapy for early rhythm control will be either by use of approved antiarrhythmic drugs (e.g. amiodarone, dronedarone, flecainide, propafenone), approved approaches and devices for ablation, or electric cardio version.
  Arms: Early rhythm control therapy
Other: Usual care for atrial fibrillation — Usual care for atrial fibrillation according to current guidelines. Usual care will mainly comprise rate control by approved drugs. We expect, that usual care will also comprise therapy for rhythm control in a small group of patients.
  Arms: Usual care

SUMMARY:
This study will determine whether early, comprehensive, rhythm control therapy prevents adverse cardiovascular outcome in patients with acute ischemic stroke and atrial fibrillation compared to usual care.

DETAILED DESCRIPTION:
trial fibrillation is the single most frequent cause of ischemic stroke and associated with a high risk of recurrent stroke and cardiovascular complications. Usual care comprises oral anticoagulation and rate control. However, it is unclear, whether early rhythm control therapy reduces the risk of recurrent stroke and cardiovascular outcomes in stroke patients with atrial fibrillation. The Early treatment of Atrial fibrillation for Stroke prevention Trial in acute STROKE (EAST-STROKE) will be an investigator-initiated, prospective, randomized, open, blinded outcome assessment (PROBE) interventional multi-center trial to test whether early, comprehensive, rhythm control therapy prevents adverse cardiovascular outcome in patients with acute ischemic stroke and atrial fibrillation compared to usual care. Primary outcome is a composite of recurrent stroke, cardiovascular death, and hospitalization due to worsening of heart failure or acute coronary syndrome. Secondary outcomes will involve a comprehensive array of clinical and safety parameters, health and socio-economic outcomes including patient reported outcome measures. In an adaptive design, up to 1,746 patients will be enrolled to demonstrate the expected treatment effect with 90% power.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke in the previous four weeks, diagnosed by imaging (CT or MRI) or clinical diagnosis
* Possibility to start the trial treatment within 4 weeks after stroke, and as soon as clinically justifiable
* AF first detected ≤1 year prior to randomization
* Informed consent

Exclusion Criteria:

* End-stage cancer or life-expectancy < 12 months due to other advanced co-morbid illness
* Prior AF ablation or surgical therapy of AF
* Patients not suitable for rhythm control of AF due to cardiac conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1746 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrent stroke, cardiovascular death, or hospitalization due to worsening of heart failure or due to acute coronary syndrome. | Through study completion, an average of 42 months
  The primary outcome measure is a composite of first recurrent stroke, cardiovascular death, and hospitalization due to worsening of heart failure or due to acute coronary syndrome as recorded by study investigators

SECONDARY OUTCOMES:
Time to first recurrent stroke | Through study completion, an average of 42 months
  Recurrent stroke as recorded by study investigators
Time to cardiovascular death | Through study completion, an average of 42 months
Time to first hospitalization due to worsening of heart failure | Through study completion, an average of 42 months
  Hospitalization due to worsening of heart failure as recorded by study investigators
Time to hospitalization due to acute coronary syndrome | Through study completion, an average of 42 months
  Hospitalization due to acute coronary syndrome as recorded by study investigators
Time to recurrent AF | Through study completion, an average of 42 months
Cardiovascular hospitalization | Through study completion, an average of 42 months
  Cardiovascular hospitalization as recorded by study investigators
All-cause hospitalizations | Through study completion, an average of 42 months
  All-cause hospitalizations as recorded by study investigators
Time in sinus rhythm | Through study completion, an average of 42 months
Functional status assessed by the modified Rankin Scale | at 12 and 24 months
  Modified Ranking Scale ranging from 0 (no symptoms) to 6 (death) with lower values indicating better status
Quality of life assessed by the EuroQol five-dimensional questionnaire (EQ-5D) | at 12 and 24 months
  The EQ-5D index will be calculated with higher values indicating better health state
Cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | at 12 and 24 months
  The MoCA ranges for 0 to 30, with higher values indicating better cognitive function
Cost of therapy | Through study completion, an average of 42 months

OTHER OUTCOMES:
All-cause mortality | Through study completion, an average of 42 months
  Death from any cause
Severe bleeding complications | Through study completion, an average of 42 months
  Intracranial hemorrhage, major bleeding
Adverse events | Through study completion, an average of 42 months
  Adverse events related to the study intervention with special emphasis on proarrhythmia and complications due to interventions

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

IPD SHARING:
Plan to Share IPD: No